CLINICAL TRIAL: NCT03795116
Title: Light Emitting Diode-Red Light (LED-RL) Phototherapy for Skin Scarring Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Principal Investigator, Jared Jagdeo, MD, MS, Associate Professor of Dermatology, State University of New York - Downstate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1304108
Record Dates: First submitted 2018-12-20; First posted 2019-01-07 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Fibrosis; Skin Scarring; Skin Wound; Hypertrophic Scar; Scar; Keloid
Keywords: Light emitting diode; Light emitting diode-red light; Visible red light; Skin fibrosis; Wound healing; Scarring
MeSH Terms: conditions — Fibrosis; Cicatrix; Cicatrix, Hypertrophic; Keloid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a single-blind study. Participants and clinicians involved in subjective efficacy assessments will be blind to the study intervention (LED-RL phototherapy versus mock therapy). The principal investigator, along with the research coordinator who administers the LED-RL phototherapy, will be aware of each participant's treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- LED-RL phototherapy (Experimental): Thirty subjects will be randomly allocated to three treatment groups to receive LED-RL phototherapy or temperature-matched mock irradiation (control) to either periauricular incision site at fluences of 160 J/cm2, 320 J/cm2, or 480 J/cm2. Starting one week after surgery (postoperative days 4-8), treatments will be administered three times weekly for three consecutive weeks.
  Interventions: Device: LED-RL phototherapy
- Mock irradiation (Sham Comparator): Thirty subjects will be randomly allocated to three treatment groups to receive LED-RL phototherapy or temperature-matched mock irradiation (control) to either periauricular incision site at fluences of 160 J/cm2, 320 J/cm2, or 480 J/cm2. Starting one week after surgery (postoperative days 4-8), treatments will be administered three times weekly for three consecutive weeks.
  Interventions: Device: Mock irradiation

INTERVENTIONS:
Device: LED-RL phototherapy — The LED-RL treatment device has a 4.7 cm x 6.1 cm rectangular array of LEDs and emits visible red light (633 nm) at a power density of 360.2 W/m2 at room temperature and a distance of 10 mm from the target surface.
  Other Names: Omnilux handheld LED system (GlobalMed Technologies, Glen Ellen, CA)
  Arms: LED-RL phototherapy
Device: Mock irradiation — The mock therapy device is designed to sound, look, and feel identical to the LED-RL treatment device (i.e., has the same physical components and thermal output), except it does not emit visible red light.
  Arms: Mock irradiation

SUMMARY:
Skin scarring (fibrosis) is a common complication in the wound healing process and remains a therapeutic challenge. Scar formation often occurs following injury to the skin such as surgery, trauma, and burns. The goal of this study is to evaluate the safety and efficacy of visible red light as a modality to reduce skin scarring after mini-facelift surgery. Based on laboratory data, light emitting diode-red light (LED-RL) phototherapy may lessen post-surgical skin fibrosis clinically.

DETAILED DESCRIPTION:
Skin fibrosis is a significant global health problem that has a profoundly negative impact on quality of life. Characterized by excessive fibroblast proliferation and collagen deposition, skin fibrosis underlies a wide spectrum of dermatologic conditions ranging from pathologic scars secondary to injury (e.g., burns, surgery, trauma) to immune-mediated diseases. Effective anti-scarring therapeutics remain an unmet need, underscoring the importance of developing novel approaches to treat and prevent skin fibrosis.

In vitro data show that LED-RL can modulate key cellular and molecular processes involved in skin fibrosis. Two phase I clinical trials (STARS 1 and STARS 2) demonstrated the safety and tolerability of LED-RL at fluences of 160 J/cm2 up to 480 J/cm2 on normal human skin. The administration of LED-RL phototherapy in the early postoperative period may optimize wound healing and prevent excessive scarring. The results from this study may change the current treatment paradigm for fibrotic skin diseases and help to pioneer LED-RL as a safe, non-invasive, cost-effective, portable, at-home therapy for scars.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent for all study procedures
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Suitable candidate for elective mini-facelift surgery
* Pass a screening photosensitivity test

Exclusion Criteria:

* Current use of any photosensitizing medications
* Light-sensitive conditions
* Diabetes mellitus
* Systemic lupus erythematosus
* Current tobacco use
* History of bleeding or coagulation disorder
* Lax skin associated with genetic disorders
* Open wounds on the face or neck
* Fibrotic skin disease, pre-existing scar(s), or other skin conditions affecting the periauricular skin
* History of surgery or procedure involving or affecting the periauricular skin within the past 6 months (e.g., prior facelift, fillers, laser therapy)
* Tattoos that cover the proposed treatment sites on the periauricular skin
* Any other medical condition(s) that could be compromised by exposure to the proposed treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen JK, Weedon J, Jakus J, Heilman E, Isseroff RR, Siegel DM, Jagdeo JR. A dose-ranging, parallel group, split-face, single-blind phase II study of light emitting diode-red light (LED-RL) for skin scarring prevention: study protocol for a randomized controlled trial. Trials. 2019 Jul 15;20(1):432. doi: 10.1186/s13063-019-3546-6. PMID 31307501

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30 participants were included in the study. This was a split-face study in which each patient received LED-RL phototherapy (i.e. low, medium, or high dose) on one preauricular incision site and mock phototherapy on the other preauricular incision site.
Units Other Than Participants: Incision Sites
Groups:
- LED-RL Phototherapy Group 1: 30 subjects were randomly allocated to three treatment groups to receive LED-RL phototherapy or temperature-matched mock irradiation (control) to either periauricular incision site at fluences of 160 J/cm2, 320 J/cm2, or 480 J/cm2. Starting one week after surgery (postoperative days 4-8), treatments will be administered three times weekly for three consecutive weeks.
  LED-RL phototherapy group 1: Received Low dose LED-RL (160 J/cm2) for 30 minutes
- Mock Irradiation Group 1: Thirty subjects will be randomly allocated to three treatment groups to receive LED-RL phototherapy or temperature-matched mock irradiation (control) to either periauricular incision site at fluences of 160 J/cm2, 320 J/cm2, or 480 J/cm2. Starting one week after surgery (postoperative days 4-8), treatments will be administered three times weekly for three consecutive weeks.
  Mock irradiation group 1: Received mock phototherapy for 30 minutes.
- LED-RL Phototherapy Group 2: 30 subjects were randomly allocated to three treatment groups to receive LED-RL phototherapy or temperature-matched mock irradiation (control) to either periauricular incision site at fluences of 160 J/cm2, 320 J/cm2, or 480 J/cm2. Starting one week after surgery (postoperative days 4-8), treatments will be administered three times weekly for three consecutive weeks.
  LED-RL phototherapy group 2: Received medium dose LED-RL (320 J/cm2) for 60 minutes
- Mock Irradiation Group 2: Thirty subjects will be randomly allocated to three treatment groups to receive LED-RL phototherapy or temperature-matched mock irradiation (control) to either periauricular incision site at fluences of 160 J/cm2, 320 J/cm2, or 480 J/cm2. Starting one week after surgery (postoperative days 4-8), treatments will be administered three times weekly for three consecutive weeks.
  Mock irradiation group 2: Received mock phototherapy for 60 minutes.
- LED-RL Phototherapy Group 3: 30 subjects were randomly allocated to three treatment groups to receive LED-RL phototherapy or temperature-matched mock irradiation (control) to either periauricular incision site at fluences of 160 J/cm2, 320 J/cm2, or 480 J/cm2. Starting one week after surgery (postoperative days 4-8), treatments will be administered three times weekly for three consecutive weeks.
  LED-RL phototherapy group 3: Received high dose LED-RL (480 J/cm2) for 90 minutes
- Mock Irradiation Group 3: Thirty subjects will be randomly allocated to three treatment groups to receive LED-RL phototherapy or temperature-matched mock irradiation (control) to either periauricular incision site at fluences of 160 J/cm2, 320 J/cm2, or 480 J/cm2. Starting one week after surgery (postoperative days 4-8), treatments will be administered three times weekly for three consecutive weeks.
  Mock irradiation group 3: Received mock phototherapy for 90 minutes.
Period: Overall Study
Arm/Group | LED-RL Phototherapy Group 1 | Mock Irradiation Group 1 | LED-RL Phototherapy Group 2 | Mock Irradiation Group 2 | LED-RL Phototherapy Group 3 | Mock Irradiation Group 3
Started | 10; 10 Incision Sites | 10; 10 Incision Sites | 10; 10 Incision Sites | 10; 10 Incision Sites | 10; 10 Incision Sites | 10; 10 Incision Sites
Completed | 6; 6 Incision Sites | 6; 6 Incision Sites | 9; 9 Incision Sites | 9; 9 Incision Sites | 9; 9 Incision Sites | 9; 9 Incision Sites
Not Completed | 4; 4 Incision Sites | 4; 4 Incision Sites | 1; 1 Incision Sites | 1; 1 Incision Sites | 1; 1 Incision Sites | 1; 1 Incision Sites

BASELINE CHARACTERISTICS:
Population: 30 participants were enrolled and included in the split-face study (i.e., began the study protocol).
Groups:
- All Participants Group 1: 30 subjects were randomly allocated to three treatment groups to receive LED-RL phototherapy or temperature-matched mock irradiation (control) to either periauricular incision site at fluences of 160 J/cm2, 320 J/cm2, or 480 J/cm2. Starting one week after surgery (postoperative days 4-8), treatments will be administered three times weekly for three consecutive weeks.
  Group 1 participants received Low dose LED-RL (160 J/cm2) for 30 minutes on one incision site and mock phototherapy for 30 minutes on the other incision site.
- All Participants Group 2: 30 subjects were randomly allocated to three treatment groups to receive LED-RL phototherapy or temperature-matched mock irradiation (control) to either periauricular incision site at fluences of 160 J/cm2, 320 J/cm2, or 480 J/cm2. Starting one week after surgery (postoperative days 4-8), treatments will be administered three times weekly for three consecutive weeks.
  Group 2 participants received medium dose LED-RL (320 J/cm2) for 60 minutes on one incision site and mock phototherapy for 60 minutes on the other incision site.
- All Participants Group 3: 30 subjects were randomly allocated to three treatment groups to receive LED-RL phototherapy or temperature-matched mock irradiation (control) to either periauricular incision site at fluences of 160 J/cm2, 320 J/cm2, or 480 J/cm2. Starting one week after surgery (postoperative days 4-8), treatments will be administered three times weekly for three consecutive weeks.
  Group 3 participants received high dose LED-RL (480 J/cm2) for 90 minutes on one incision site and mock phototherapy for 90 minutes on the other incision site.
- Total: Total of all reporting groups
Arm/Group | All Participants Group 1 | All Participants Group 2 | All Participants Group 3 | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (8.2) | 52.4 (7.2) | 56.3 (7.4) | 54.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 30
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White non-hispanic | 5 | 6 | 8 | 19
  White hispanic | 2 | 3 | 1 | 6
  Black or African American | 2 | 1 | 1 | 4
  Two or more races | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Scar Pliability Between the Treated and Control Incision Sites as Measured by Skin Elasticity at 6 Months Compared to Baseline
Description: The ElastiMeter, a non-invasive indentation instrument, will be used to evaluate skin elasticity (i.e., skin stiffness) of the LED-RL-treated scar versus the untreated scar. Skin elasticity is measured in Newtons/meters (N/m).
Time Frame: 1 month, 3 months, 6 months
Population: Collected data were not considered valid due to an equipment malfunction.
Arm/Group | LED-RL Phototherapy | Mock Irradiation
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Scar Pliability Between the Treated and Control Incision Sites as Measured by Skin Induration at Three Follow-up Time Points Compared to Baseline
Description: The SkinFibroMeter, a non-invasive indentation instrument, will be used to evaluate the induration of the skin and subcutaneous tissue (i.e., hardness) of the LED-RL-treated scar versus the untreated scar. Skin induration is measured in Newtons (N).
Time Frame: Baseline assessment was completed on post-operative day 5, before LED-RL or mock phototherapy treatment. Follow-up visits were scheduled on approximately post-operative day 30 (1 month), post-operative 90 (3 months), and post-operative day 180 (6 months).
Population: In this split-face study, 10 subjects were randomly assigned to each LED-RL group (low, medium, or high dose). While 30 subjects participated in the study, there were 60 total preauricular incision sites (in each participant, one site treated with LED-RL and the other with mock phototherapy). Due to subjects missing assessment visits (i.e. personal reasons, withdrawals, etc), there may be less than 10 subjects per group analyzed at each time point.
Measure: Median (Inter-Quartile Range); unit: Newton
Units Other Than Participants: Incision Sites
Arm/Group | LED-RL Phototherapy Group 1 | Mock Irradiation Group 1 | LED-RL Phototherapy Group 2 | Mock Irradiation Group 2 | LED-RL Phototherapy Group 3 | Mock Irradiation Group 3
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Number analyzed (Incision Sites) | 10 | 10 | 10 | 10 | 10 | 10
Newton
  Baseline | .08 [.04 to .14] | .05 [.02 to .08] | .09 [.03 to .13] | .06 [.04 to .08] | .06 [.04 to .07] | .07 [.02 to .08]
  1 month: number analyzed (Participants) | 9 | 9 | 10 | 10 | 9 | 9
  1 month: number analyzed (Incision Sites) | 9 | 9 | 10 | 10 | 9 | 10
  1 month | .05 [.04 to .08] | .04 [.03 to .08] | .06 [.04 to .08] | .05 [.03 to .12] | .05 [.03 to .08] | .04 [.02 to .04]
  3 months: number analyzed (Participants) | 8 | 8 | 9 | 9 | 10 | 10
  3 months: number analyzed (Incision Sites) | 8 | 8 | 9 | 9 | 10 | 10
  3 months | .03 [.03 to .06] | .04 [.02 to .05] | .04 [.03 to .07] | .04 [.04 to .07] | .05 [.04 to .06] | .06 [.04 to .08]
  6 months: number analyzed (Participants) | 6 | 6 | 9 | 9 | 9 | 9
  6 months: number analyzed (Incision Sites) | 6 | 6 | 9 | 9 | 9 | 9
  6 months | .03 [.02 to .03] | .03 [.02 to .03] | .02 [.02 to .03] | .03 [.03 to .03] | .03 [.02 to .03] | .02 [.02 to .03]

3. Secondary Outcome: Observer Scar Assessment Scale
Description: The scale consists of six items rated from 1 to 10, where 1 is "normal skin" and 10 is the "worst imaginable scar". The observer (i.e., investigator) evaluates scar vascularity, pigmentation, thickness, relief, pliability, and surface area. The scores of each of the six items are summed for a total score (range 6 to 60).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Units Other Than Participants: Incision Sites
Arm/Group | LED-RL Phototherapy Group 1 | Mock Irradiation Group 1 | LED-RL Phototherapy Group 2 | Mock Irradiation Group 2 | LED-RL Phototherapy Group 3 | Mock Irradiation Group 3
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Number analyzed (Incision Sites) | 10 | 10 | 10 | 10 | 10 | 10
score on a scale
  Baseline | 16.5 [14.0 to 20.0] | 16.5 [15.0 to 21.0] | 19.0 [16.0 to 21.0] | 14.0 [13.0 to 17.0] | 18.0 [16.0 to 19.0] | 16.5 [15.0 to 20.0]
  1 month: number analyzed (Participants) | 9 | 9 | 10 | 10 | 9 | 9
  1 month: number analyzed (Incision Sites) | 9 | 9 | 10 | 10 | 9 | 9
  1 month | 17.0 [15.0 to 18.0] | 17.0 [14.0 to 19.0] | 13.0 [11.0 to 16.0] | 17.5 [11.0 to 19.0] | 19.0 [17.0 to 21.0] | 13.0 [12.0 to 15.0]
  3 months: number analyzed (Participants) | 8 | 8 | 9 | 9 | 10 | 10
  3 months: number analyzed (Incision Sites) | 8 | 8 | 9 | 9 | 10 | 10
  3 months | 12.5 [11.5 to 17.0] | 15.0 [14.0 to 16.0] | 12.0 [11.0 to 18.0] | 14.0 [9.0 to 18.0] | 15.0 [12.0 to 19.0] | 13.0 [12.0 to 14.0]
  6 months: number analyzed (Participants) | 6 | 6 | 9 | 9 | 9 | 9
  6 months: number analyzed (Incision Sites) | 6 | 6 | 9 | 9 | 9 | 9
  6 months | 9.0 [8.0 to 18.0] | 12.5 [11.0 to 14.0] | 8.0 [8.0 to 20.0] | 14.0 [12.0 to 16.0] | 13.0 [10.0 to 15.0] | 12.0 [8.0 to 19.0]

4. Secondary Outcome: Visual Analog Scale (VAS) Scoring of Digital Photographs of Scars
Description: The scar images will be rated by two independent, blinded dermatologists using a VAS. The VAS is presented as a 10 cm horizontal line, where the extreme ends of 0 indicates "normal skin" and 10 corresponds to the "worst possible scar," for each of the following scar attributes: pigmentation, vascularity, observer comfort, contour, and overall severity.
Time Frame: as for outcome 2
Population: Data were not collected for this outcome measure.
Arm/Group | LED-RL Phototherapy | Mock Irradiation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Dermal Collagen Concentration
Description: A non-invasive, handheld diffuse reflectance probe will be used to measure collagen concentration in the dermis at each incision site. The scale ranges from 10 to 99 and the collagen measurement corresponds to the half of the optical scattering coefficient of the dermis.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Units Other Than Participants: Incision Sites
Arm/Group | LED-RL Phototherapy Group 1 | Mock Irradiation Group 1 | LED-RL Phototherapy Group 2 | Mock Irradiation Group 2 | LED-RL Phototherapy Group 3 | Mock Irradiation Group 3
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Number analyzed (Incision Sites) | 10 | 10 | 10 | 10 | 10 | 10
arbitrary units
  Baseline | 48.7 [41.0 to 59.5] | 52.0 [37.0 to 62.6] | 51.0 [34.0 to 59.0] | 50.5 [42.0 to 62.0] | 47.7 [39.3 to 62.0] | 52.5 [46.0 to 62.0]
  1 month: number analyzed (Participants) | 9 | 9 | 10 | 10 | 9 | 9
  1 month: number analyzed (Incision Sites) | 9 | 9 | 10 | 10 | 9 | 9
  1 month | 60.3 [50.0 to 62.0] | 47.0 [29.3 to 56.3] | 50.7 [44.7 to 58.0] | 55.2 [43.7 to 60.0] | 52.7 [42.3 to 60.7] | 57.0 [48.3 to 60.3]
  3 months: number analyzed (Participants) | 8 | 8 | 9 | 9 | 10 | 10
  3 months: number analyzed (Incision Sites) | 8 | 8 | 9 | 9 | 10 | 10
  3 months | 57.5 [47.8 to 60.3] | 57.4 [55.5 to 61.5] | 58.3 [55.0 to 60.7] | 57.3 [54.7 to 58.0] | 58.7 [48.0 to 59.6] | 58.7 [55.6 to 62.0]
  6 months: number analyzed (Participants) | 6 | 6 | 9 | 9 | 9 | 9
  6 months: number analyzed (Incision Sites) | 6 | 6 | 9 | 9 | 9 | 9
  6 months | 57.0 [55.3 to 58.7] | 56.5 [53.0 to 60.3] | 60.0 [56.0 to 61.7] | 61.0 [54.7 to 61.3] | 56.7 [50.3 to 57.0] | 59.3 [56.7 to 61.3]

6. Secondary Outcome: Dermal Water Concentration
Description: A non-invasive, handheld diffuse reflectance probe will be used to measure water concentration in the dermis at each incision site. Infrared light is emitted at different wavelengths to retrieve the scattering and the absorption coefficients of the dermis. The more water, the less reflectance. Concentration ranges from 40% to 85%.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage
Units Other Than Participants: Incision Sites
Arm/Group | LED-RL Phototherapy Group 1 | Mock Irradiation Group 1 | LED-RL Phototherapy Group 2 | Mock Irradiation Group 2 | LED-RL Phototherapy Group 3 | Mock Irradiation Group 3
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Number analyzed (Incision Sites) | 10 | 10 | 10 | 10 | 10 | 10
percentage
  Baseline | 63.0 [60.0 to 64.3] | 65.3 [62.3 to 66.0] | 60.7 [58.7 to 62.0] | 62.7 [60.0 to 66.0] | 63.2 [62.0 to 67.7] | 66.2 [63.0 to 68.0]
  1 month: number analyzed (Participants) | 9 | 9 | 10 | 10 | 9 | 9
  1 month: number analyzed (Incision Sites) | 9 | 9 | 10 | 10 | 9 | 9
  1 month | 64.0 [62.0 to 65.0] | 62.3 [61.3 to 63.3] | 60.2 [58.3 to 61.7] | 62.3 [58.3 to 63.3] | 60.6 [58.7 to 62.7] | 64.0 [60.0 to 65.0]
  3 months: number analyzed (Participants) | 8 | 8 | 9 | 9 | 10 | 10
  3 months: number analyzed (Incision Sites) | 8 | 8 | 9 | 9 | 10 | 10
  3 months | 63.0 [59.7 to 67.8] | 61.4 [59.0 to 67.3] | 63.0 [59.7 to 66.3] | 60.7 [59.3 to 62.3] | 61.7 [60.6 to 63.3] | 62.0 [57.0 to 67.6]
  6 months: number analyzed (Participants) | 6 | 6 | 9 | 9 | 9 | 9
  6 months: number analyzed (Incision Sites) | 6 | 6 | 9 | 9 | 9 | 9
  6 months | 62.5 [59.0 to 64.3] | 61.2 [59.7 to 64.0] | 63.7 [62.3 to 68.3] | 63.0 [62.7 to 64.7] | 62.0 [61.3 to 62.3] | 64.0 [61.3 to 64.7]

7. Secondary Outcome: 3D Imaging Analysis: Pigmentation of Scar Tissue
Description: A 3D digital imaging system will be used to construct 3D images of the scars for colorimetric analyses, including quantitative measurements of pigmentation at each incision site.
Time Frame: as for outcome 2
Population: Data were not collected for this outcome measure.
Arm/Group | LED-RL Phototherapy | Mock Irradiation
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: 3D Imaging Analysis: Vascularity of Scar Tissue
Description: A 3D digital imaging system will be used to construct 3D images of the scars for colorimetric analyses, including quantitative measurements of vascularity at each incision site.
Time Frame: as for outcome 2
Population: Data were not collected for this outcome measure.
Arm/Group | LED-RL Phototherapy | Mock Irradiation
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: 3D Imaging Analysis: Volume of Elevation of Scar Tissue
Description: A 3D digital imaging system will be used to construct 3D images of the scars for skin profilometry analyses, including quantitative measurements of tissue volume at each incision site.
Time Frame: as for outcome 2
Population: Data were not collected for this outcome measure.
Arm/Group | LED-RL Phototherapy | Mock Irradiation
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Histological Analysis: Collagen Content of Scar Tissue (Optional)
Description: The histological changes that occur in vivo in response to LED-RL phototherapy will be evaluated by examination of pre- and post-treated skin tissue. Skin specimens will be obtained via optional 2 mm punch biopsy and stained for collagen fibers.
Time Frame: Skin specimens will be obtained via optional 2 mm punch biopsy on post-operative day 0 (prior to surgery) and post-operative day 30 (first follow-up visit after completion of LED-RL treatment).
Population: Biopsy was optional. This outcome measure was not performed for any subjects.
Arm/Group | LED-RL Phototherapy | Mock Irradiation
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Participants Experiencing Adverse Events in Each Treatment Group
Description: Subjects will be provided with a daily diary to record any adverse events experienced during the three-week intervention period. Treatment sessions will be monitored closely for the occurrence of any safety issues or adverse events, as reported by the subject or observed by the clinical research team. At each follow up visit, patients will be asked about adverse effects.
Time Frame: From first LED-RL and mock phototherapy treatment session on post-operative day 5 until final follow-up visit on post-operative day 180 (6 month follow-up).
Population: This was a split-face study including 30 participants. Each participant received LED-RL phototherapy (i.e. low, medium, or high dose) on one preauricular incision site and mock phototherapy on the other preauricular incision site.
Measure: Count of Participants; unit: Participants
Groups:
- Mock Irradiation Group 1: 30 subjects will be randomly allocated to three treatment groups to receive LED-RL phototherapy or temperature-matched mock irradiation (control) to either periauricular incision site at fluences of 160 J/cm2, 320 J/cm2, or 480 J/cm2. Starting one week after surgery (postoperative days 4-8), treatments will be administered three times weekly for three consecutive weeks.
  Mock irradiation group 1: Received mock phototherapy for 30 minutes.
- Mock Irradiation Group 2: 30 subjects will be randomly allocated to three treatment groups to receive LED-RL phototherapy or temperature-matched mock irradiation (control) to either periauricular incision site at fluences of 160 J/cm2, 320 J/cm2, or 480 J/cm2. Starting one week after surgery (postoperative days 4-8), treatments will be administered three times weekly for three consecutive weeks.
  Mock irradiation group 2: Received mock phototherapy for 60 minutes.
Arm/Group | LED-RL Phototherapy Group 1 | Mock Irradiation Group 1 | LED-RL Phototherapy Group 2 | Mock Irradiation Group 2 | LED-RL Phototherapy Group 3 | Mock Irradiation Group 3
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Participants
  localized bulla | 0 | 0 | 1 | 0 | 1 | 0
  localized facial swelling | 0 | 0 | 0 | 0 | 1 | 0
  no adverse events | 10 | 10 | 9 | 10 | 8 | 10

12. Secondary Outcome: Patient Scar Assessment Scale
Description: The scale consists of six items rated from 1 to 10, where 1 is "normal skin" and 10 is the "worst imaginable scar". The patient assesses pain, itching, color, stiffness, thickness, and irregularity. The scores of each of the six items are summed for a total score (range 6 to 60).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Units Other Than Participants: Incision Sites
Arm/Group | LED-RL Phototherapy Group 1 | Mock Irradiation Group 1 | LED-RL Phototherapy Group 2 | Mock Irradiation Group 2 | LED-RL Phototherapy Group 3 | Mock Irradiation Group 3
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Number analyzed (Incision Sites) | 10 | 10 | 10 | 10 | 10 | 10
score on a scale
  Baseline | 36.0 [27.0 to 42.0] | 37.0 [24.0 to 41.0] | 32.0 [23.0 to 34.0] | 30.5 [27.0 to 32.0] | 26.5 [21.0 to 33.0] | 28.5 [24.0 to 48.0]
  1 month: number analyzed (Participants) | 9 | 9 | 10 | 10 | 9 | 9
  1 month: number analyzed (Incision Sites) | 9 | 9 | 10 | 10 | 9 | 9
  1 month | 25.0 [21.0 to 34.0] | 25.0 [19.0 to 34.0] | 24.0 [19.0 to 29.0] | 23.5 [18.0 to 30.0] | 17.0 [13.0 to 37.0] | 26.0 [13.0 to 37.0]
  3 months: number analyzed (Participants) | 8 | 8 | 9 | 9 | 10 | 10
  3 months: number analyzed (Incision Sites) | 8 | 8 | 9 | 9 | 10 | 10
  3 months | 12.5 [12.0 to 18.0] | 15.0 [12.0 to 25.5] | 18.0 [17.0 to 26.0] | 21.0 [18.0 to 26.0] | 17.5 [14.0 to 32.0] | 20.0 [12.0 to 26.0]
  6 months: number analyzed (Participants) | 6 | 6 | 9 | 9 | 9 | 9
  6 months: number analyzed (Incision Sites) | 6 | 6 | 9 | 9 | 9 | 9
  6 months | 12.0 [7.0 to 17.0] | 10.5 [10.0 to 12.0] | 23.0 [12.0 to 28.0] | 18.0 [16.0 to 24.0] | 13.0 [10.0 to 25.0] | 17.0 [11.0 to 26.0]

ADVERSE EVENTS:
Time Frame: LED-RL and mock phototherapy treatment sessions were monitored for the occurrence of safety concerns and AEs, as reported by the patient or observed by the research team. Patients recorded AEs during the three-week LED-RL and mock phototherapy treatment period in a home diary. At each visit, participants were asked about AEs.
Arm/Group | LED-RL Phototherapy Group 1 | Mock Irradiation Group 1 | LED-RL Phototherapy Group 2 | Mock Irradiation Group 2 | LED-RL Phototherapy Group 3 | Mock Irradiation Group 3
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 1/10 | 0/10 | 2/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LED-RL Phototherapy Group 1 (N=10) | Mock Irradiation Group 1 (N=10) | LED-RL Phototherapy Group 2 (N=10) | Mock Irradiation Group 2 (N=10) | LED-RL Phototherapy Group 3 (N=10) | Mock Irradiation Group 3 (N=10)
Localized Bulla (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Localized Facial Swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT03795116/Prot_SAP_000.pdf